CLINICAL TRIAL: NCT03096470
Title: Clinical Analysis of Two Methods for Closed Reduction of Developmental Dislocation of the Hip by Prolonged Traction < 6 Months----An Multicenter Prospective Observational Study
Brief Title: Closed Reduction With Anesthesia and no Anesthesia for Developmental Dislocation of the Hip < 6 Months
Status: Completed | Type: Observational
Sponsor: The Fuzhou No 2 Hospital (Other)
Responsible Party: Principal Investigator, Shunyou Chen, Director,Orthopaedics, The Fuzhou No 2 Hospital
Other Study IDs: SChen1
Record Dates: First submitted 2017-03-10; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Developmental Dislocation of the Hip; Reduction Deformity of Limb
MeSH Terms: conditions — Ectromelia | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anesthesia: The children were treated with closed reduction with anesthesia after prolonged traction
  Interventions: Procedure: anesthesia
- No anesthesia: The children were treated with closed reduction with no anesthesia after prolonged traction
  Interventions: Procedure: anesthesia

INTERVENTIONS:
Procedure: anesthesia — no anesthesia

SUMMARY:
The purpose of this study is to compare the efficacy of closed reduction with anesthesia and no anesthesia for developmental dislocation of the hip < 6 months

DETAILED DESCRIPTION:
We treated children (<6 months) with prolonged traction before an attempted closed reduction. And compare the efficacy of closed reduction with anesthesia and no anesthesia for developmental dislocation of the hip. All the patients were followed up for a minimum of 18 months in order to identify any avascular changes in the femoral head. The presence of avascular necrosis was assessed by the criteria of Salter.

ELIGIBILITY:
Inclusion Criteria:

* The patients with GrafⅢ/Ⅳtype DDH diagnosed by ultrasound or if they were IHDI (International Hip Dysplasia Institute) grade III or IV on radiographs，and The infants who were <6 months of age. Patients were followed for at least 18 months,by which time they had either completed treatment with no evidence of requiring further treatment or were treated surgically after failing brace treatment.

Exclusion Criteria:

* Infants were excluded if they had multiple congenital abnormalities, had prior treatment in other centres, or showed teratological dislocations. The last were defined as fixed dislocation of the hip in association with either a recognised syndrome or a neurological disorder.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: developmental dislocation of the hip（ < 6 months）
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Successful treatment | Through study completion, an average of 2 year.
  obtain and maintain reduction of the hip following bracing with no subsequent surgical treatment

SECONDARY OUTCOMES:
Radiographic evaluation | Through study completion, an average of 2 year.
  Radiographic data collected included evaluation of the Shenton line, the acetabular index, the IHDI grade, the state of ossification of the femoral head, a description of the teardrop, the lateral center-edge angle, and the presence of osteonecrosis of the femoral head

OTHER OUTCOMES:
The complication | Through study completion, an average of 2 year.
  the presence of osteonecrosis of the femoral head， Avascular necrosis was assessed using the criteria of Salter

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cashman JP, Round J, Taylor G, Clarke NM. The natural history of developmental dysplasia of the hip after early supervised treatment in the Pavlik harness. A prospective, longitudinal follow-up. J Bone Joint Surg Br. 2002 Apr;84(3):418-25. doi: 10.1302/0301-620x.84b3.12230. PMID 12002504
- [Background] Upasani VV, Bomar JD, Matheney TH, Sankar WN, Mulpuri K, Price CT, Moseley CF, Kelley SP, Narayanan U, Clarke NM, Wedge JH, Castaneda P, Kasser JR, Foster BK, Herrera-Soto JA, Cundy PJ, Williams N, Mubarak SJ. Evaluation of Brace Treatment for Infant Hip Dislocation in a Prospective Cohort: Defining the Success Rate and Variables Associated with Failure. J Bone Joint Surg Am. 2016 Jul 20;98(14):1215-21. doi: 10.2106/JBJS.15.01018. PMID 27440570
- [Background] Fukiage K, Futami T, Ogi Y, Harada Y, Shimozono F, Kashiwagi N, Takase T, Suzuki S. Ultrasound-guided gradual reduction using flexion and abduction continuous traction for developmental dysplasia of the hip: a new method of treatment. Bone Joint J. 2015 Mar;97-B(3):405-11. doi: 10.1302/0301-620X.97B3.34287. PMID 25737526
- [Background] Yamada N, Maeda S, Fujii G, Kita A, Funayama K, Kokubun S. Closed reduction of developmental dislocation of the hip by prolonged traction. J Bone Joint Surg Br. 2003 Nov;85(8):1173-7. doi: 10.1302/0301-620x.85b8.14208. PMID 14653603